CLINICAL TRIAL: NCT07083245
Title: Coda Comfort Crew Pilot Project: Assessing and Addressing the Psychosocial Needs of Chemotherapy Patients With the Gatineau Cancer Center
Acronym: CCC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coda Foundation (Other)
Responsible Party: Principal Investigator, Patrick Shaw, Medical Student, Coda Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: codacomfortcrewpilotstudy
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Cancer
Keywords: Cancer; Psychosocial; Anxiety; Depression; distress
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychosocial support group (Experimental): This arm will receive treatment through the form of the Coda Comfort Crews intervention, including material and psychosocial support. This will be done through material gifts, watching movies and playing board games as well as conversations together during chemotherapy treatments.
  Interventions: Behavioral: Psychosocial care

INTERVENTIONS:
Behavioral: Psychosocial care — Psychosocial support to chemotherapy patients during their treatment sessions through conversations, board games, movies, and gift baskets

SUMMARY:
This study seeks to examine the impact of a psychosocial intervention offered by the Coda Comfort Crew, which entails providing conversational support, parallel play, material support through gift bags and more on anxiety and depression, and on distress experienced by patients undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years old)
* Diagnosed with cancer and undergoing chemotherapy at the Gatineau Cancer Center during the intervention and study period
* Able to understand and provide informed consent
* Sufficient understanding of French or English

Exclusion Criteria:

* Major cognitive impairment preventing understanding
* Severe medical or psychiatric comorbidities limiting participation
* Minors (< 18 years old)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Distress | 3 months
  A checklist of things that might evoke unpleasant experiences of a mental, physical, social, or spiritual nature, as well as a 1-10 scale of overall distress.
HADS | 3 months
  Hospital anxiety and depression scale scores

IPD SHARING:
Plan to Share IPD: No